CLINICAL TRIAL: NCT06763484
Title: Paroxetine Versus Placebo for Vasomotor Symptom Management in Surgical Menopause. Randomized Double-blind Clinical Trial
Brief Title: Paroxetine Versus Placebo for Vasomotor Symptom Management in Surgical Menopause
Acronym: MENOXTINA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGO-UNAH-48-2-2025
Record Dates: First submitted 2024-12-30; First posted 2025-01-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Menopause Syndrome; Menopause Surgical; Hot Flashes
Keywords: Menopause Syndrome; Menopause Surgical; Hot Flashes; Paroxetine
MeSH Terms: conditions — Hot Flashes | interventions — Paroxetine; Starch

STUDY DESIGN:
Intervention Model Description: parallel-group, efficacy, superiority, double-blind clinical trial
Who Masked: Participant, Investigator
Masking Description: To eliminate researcher bias, a third research participant will place the capsules containing the soy isoflavonate in one bottle and the placebo in another bottle. The bottles will be labeled as group A and group B, but the researchers will not know which is in which group, to ensure that the study intervention and the control/placebo are as indistinguishable as possible to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paroxetine (Experimental): 20mg Paroxetine once daily for 12 weeks
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): 1 placebo capsule containing starch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Paroxetine — 20 mg PO daily
  Arms: Paroxetine
Dietary Supplement: Placebo — 1 capsule starch
  Other Names: Starch
  Arms: Placebo

SUMMARY:
evaluate the efficacy of paroxetine in the management of vasomotor symptoms in patients with surgical menopause, in order to seek an alternative therapy to hormone therapy, which is associated with proinflammatory and procoagulant effects that increase the risk of thrombosis and is therefore contraindicated in people with diabetes mellitus, chronic arterial hypertension and patients with a history of thromboembolism

DETAILED DESCRIPTION:
Vasomotor symptoms that occur in the peri-menopausal and postmenopausal period are experienced by 80% of women and can greatly affect the quality of life by temporarily interrupting daily activities. These symptoms are experienced early in our study population who are induced to early menopause by undergoing surgical procedures such as total abdominal hysterectomy plus bilateral salpingo-oophorectomy.

Due to the controversy that exists about the use of hormone replacement therapy, in recent years different alternative therapies have been proposed for the management of these symptoms, mainly for those patients who have contraindications for hormone therapy. For this reason, the use of non-hormonal therapy has been investigated.

Since there are women who have contraindications to conventional therapy such as patients with cardiovascular and thrombosis risks, there is a need to search for new alternative therapies such as selective serotonin reuptake inhibitors, specifically paroxetine, so with our study we seek to evaluate how effective paroxetine is in reducing vasomotor symptoms and thus provide an alternative to this type of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical menopause attending IHSS outpatient clinic.
* Patients with surgical menopause with presence of hot flashes and night sweats.
* Surgical menopausal patients with episodes of anxiety and palpitations.
* Patients with surgical menopause who receive treatment for 6 months with Paroxetine.
* Patients who after reading and explanation of the Informed Consent agree to participate voluntarily.

Exclusion Criteria:

* Patients medicated with psychotropic drugs, including all sedatives and hypnotics.
* Patients under treatment with Menopausal Hormone Therapy.
* Patients with impaired hepatic or renal function.
* Patients with unstable heart disease.
* Patients with a history of self-destructive behaviors.
* Patients with a history of clinical diagnosis or treatment for depression or any other psychiatric disorder (including substance abuse or alcohol disorders) and any other ongoing medical condition.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Score (MRS) | Since intervention until 12 weeks
  change in the Menopause Rating Scale (MRS), which measures 11 variables with a score of 0 to 4, with 0 being the absence of symptoms, scores range from 0 to 44.

SECONDARY OUTCOMES:
Frequency of vasomotor symptoms | Since intervention until 12 weeks
  Changes in the frequency of vasomotor symptoms, The incidence of vasomotor symptoms will be assessed at each visit
side effects | Since intervention until 12 weeks
  incidence of side effects of paroxetine

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Instituto Hondureño de Seguridad Social, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Iyer TK, Fiffick AN, Batur P. Nonhormone therapies for vasomotor symptom management. Cleve Clin J Med. 2024 Apr 1;91(4):237-244. doi: 10.3949/ccjm.91a.23067. PMID 38561208